CLINICAL TRIAL: NCT03430076
Title: Polytetrafluoroethylen (PTFE) Vascular Prostheses With Heparin Bonded Luminal Surfaces vs Crude ePTFE in the Treatment of Critical Limb Ischemia Lesions in the Absence of a Suitable Autologous Vein
Brief Title: Polytetrafluoroethylen (PTFE) Vascular Prostheses With Heparin Bonded Luminal Surfaces vs Crude ePTFE
Acronym: REPLACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RC17_0205
Record Dates: First submitted 2018-01-16; First posted 2018-02-12 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Ischemia Lesions
Keywords: vascular prostheses; heparin; ischemia lesions; vascular; critical limb ischemia lesions

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Revascularization by (Propaten)® (Experimental): Revascularization by PTFE with heparin bonded luminal surface (Propaten)®
  Interventions: Procedure: revascularization; Device: Propaten®
- Revascularization by Crude PTFE (Active Comparator)
  Interventions: Procedure: revascularization; Device: Crude PTFE

INTERVENTIONS:
Procedure: revascularization — open revascularization for below-knee popliteal in the absence of an suitable autologous vein with PTFE.
Device: Propaten® — Propaten®
  Arms: Revascularization by (Propaten)®
Device: Crude PTFE — Crude PTFE
  Arms: Revascularization by Crude PTFE

SUMMARY:
Open repair could be recommended in a first line of treatment to revascularize critical limb ischemia patients or performed in a second line of treatment in case of failure of endovascular repair. A good quality vein is one of the main factors that influence the clinical success of open revascularization for below-knee popliteal. In the absence of an suitable autologous vein, prosthesis such as polytetrafluoroethylen (PTFE) graft could be an option but demonstrated worse clinical and morphological results compared to autologous greater saphenous vein. Consequently, there is still a room for improvement in CLI patients in the absence of an suitable autologous vein in whom endovascular repair failed.

Recently, PTFE with heparin-bound to the luminal surface (Hb-PTFE) significantly reduced the overall risk of primary graft failure by 37%, in particular, risk reduction was 50% in femoropopliteal bypass cases in cases with critical ischemia (58% Primary patency for crude ePTFE versus 80% primary patency for PROPATEN at 1 year follow-up) (Lindholt, et. al. 2011).

Additionally, a weighted average from the literature suggests a 76% primary patency for below knee bypasses performed with PROPATEN at one year follow-up, whereas a published meta-analysis suggests a 59% primary patency for below knee crude ePTFE at one year follow-up. At two year follow-up using the same approach, the average primary patency for PROPATEN was 67% versus 43% for standard ePTFE.

The aim of this study is to assess PTFE with heparin-bound to the luminal surface as an alternative to crude PTFE in absence of good venous conduit in patients with CLI.

DETAILED DESCRIPTION:
Patient inclusion in this study will be proposed 60 to 1-days period preceding the surgical procedure. The patient will be randomized in the crude PTFE or in the Propaten groups. Regarding the intervention, the technique used during the therapeutic procedure shall be left to the operator's discretion, except the type of the graft. Demographic, intraoperative and postoperative data will be collected prospectively. Patient will be assessed and followed up according a current care. The cost difference between both groups will be identified.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥18 years
* Patient presented critical limb ischemia (Rutherford classification: 4-6)
* Indication of below the knee bypass with an artificial graft
* Absence of an suitable autologous vein
* Patient is affiliated to the Social Security or equivalent system
* Patient has been informed of the nature of the study, agrees to its provisions and has signed the informed consent form prior to any study related procedure
* Patient agrees to undergo all protocol required follow-up examinations and requirements at the investigational site

Exclusion Criteria:

* No atheromatous disease
* Female of child bearing potential
* Patient has a history of coagulopathy or will refuse blood transfusions
* Patient is receiving or scheduled to receive anticancer therapy for malignancy within 1 year prior to or after the procedure
* Severe concomitant disease with life expectation < one year
* Known allergy to heparin
* Indication for ipsilateral major amputation
* Patient is not able to give informed consent
* Patient is currently participating in an investigational drug or device study that has not completed the primary endpoint or that clinically interferes with the current study endpoints Note: Trials requiring extended follow-up for products that were investigational, but have become commercially suitable since then, are not considered investigational trials
* In the Investigator's opinion patient has (a) co-morbid condition(s) that could limit the patient's ability to participate in the study, compliance with follow-up requirements or impact the scientific integrity of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2018-02-13 (Actual); Primary Completion 2024-01-29 (Actual); Study Completion 2024-01-29 (Actual)

PRIMARY OUTCOMES:
Primary patency at 1 year: | 1 year
  It was defined as a patent graft without any intervention to open up or prevent a graft occlusion. Demonstrably patent graft should be by a duplex ultrasound color-flow scan.

SECONDARY OUTCOMES:
Technical success defined as a patent bypass without stenosis of the proximal and the distal anastomoses. | 2 years
  Stenosis was defined as >30% diameter stenosis noted on intraoperative arteriography.
Perioperative complications | 2 years
  defined as any general complications or local complications that caused or prolonged hospitalization and/or re-intervention, lymphorrhea of more than 3-days and post-operative paresthesia that required drugs. The general complications included death from any cause, MACE. Local complications included MALE, hematoma, active bleeding, local infection, thrombosis, delayed wound healing and false aneurysm
Primary sustained clinical improvement | 1, 12 and 24 months post procedure
  defined as a wound healing and rest pain resolution for patients in CLI, without the need for repeated graft it self or anastomoses in surviving patients.
Secondary sustained clinical improvement | 1, 12 and 24 months post procedure
  defined as primary sustained clinical improvement including the need for repeated graft it self or anastomoses.
Primary patency | 1 and 24 months post procedure
  defined as a patent graft without any intervention to open up or prevent a graft occlusion. Demonstrably patent graft should be by a duplex ultrasound color-flow scan.
Major adverse cardiovascular events | 1, 12 and 24 months post procedure
  defined as MACEs including all cardiac deaths, Q wave infarction, stroke
MALE (Major Adverse Limb Event)-free survival rates in subjects with CLI randomized to Propaten vs. crude ePTFE. | 1, 6, 12 and 24 months
  MALE is defined as above-ankle amputation of the index limb or major reintervention (new bypass graft, jump/interposition graft revision, or thrombectomy/ thrombolysis).
Limb salvage defined as freedom from above-ankle amputation of the index limb | 1, 12 and 24 months post procedure
Secondary patency | 1, 12 and 24 months post procedure
  secondary patency in which graft patency is lost (occlusion) and restored by thrombectomy, thrombolysis, or transluminal angioplasty, and/or any problems with the graft itself or one of its anastomoses require revision or reconstruction. Demonstrably patent graft should be by a duplex ultrasound color-flow scan.
Assisted patency | 1, 12 and 24 months post procedure
  : Assisted patency at 1, 12 and 24 months post procedure, in which patency was never lost but maintained by prophylactic intervention. Demonstrably patent graft should be by a duplex ultrasound color-flow scan.
Death | 1, 12 and 24 months post procedure
  Death (all cause)
Ankle brachial index | 1, 6, 12 and 24 months post procedure
  Post-operative assessment (clinical, morphological, hemodynamic criteria)
Quality of life at inclusion, . | 1, 3, 6, 9, 12, 15, 18 and 24 months
  assessed according the EQ-5D-3L questionnaire
Cost utility analysis (CUA) | 2 years
  In CUA, the outcomes of an intervention are evaluated in terms of Quality-Adjusted Life-Years (QALYs). QALYs are a numerical index that encompasses both the length of life and the health-related quality-of-life.
cost-effectiveness analysis (CEA) | 2 years
  The Measure of outcome for CEA will be the number of Life Years Gained (LYG) at 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Yann Gouëffic, Pr, Principal Investigator — Saint Joseph Hospital Paris
Locations (21):
- France (21):
  - Angers University Hospital, Angers
  - Besançon University Hospital, Besançon
  - Bordeaux University Hospital - Hôpital Pellegrin, Bordeaux
  - Ambroise Paré university Hospital, Boulogne-Billancourt
  - Brest University Hospital, Brest
  - Clermont-Ferrand University Hospital, Clermont-Ferrand
  - Dijon University Hospital, Dijon
  - Lille University Hospital, Lille
  - Lyon University Hospital - Hopital Edouard Herriot, Lyon
  - Timone hospital, Marseille
  - Nancy University Hospital, Nancy
  - Nantes University Hospital, Nantes
  - Hopital Pasteur, Nice
  - Saint Joseph Hospital, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Bichat Hospital, Paris
  - Poitiers University Hospital, Poitiers
  - Reims university Hospital, Reims
  - Saint Etienne University Hospital, Saint-Etienne
  - Nouvel Hopital Civil, Strasbourg
  - Valenciennes University Hospital, Valenciennes

IPD SHARING:
Plan to Share IPD: No